CLINICAL TRIAL: NCT03708679
Title: Are Menstruel Cycle Phases Effective on Preoperative Anxiety? Prospective, Clinical Study
Brief Title: Effects of Menstrual Cycle on Preoperative Anxiety
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assist. Prof, Yuzuncu Yil University
Other Study IDs: Menstruel Cycle Anxiety
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Menstrual Cycle; Perioperative Hypertension; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group F: Patients with menstrual cycle between 8-12 days were called Group F (Follicular phase)
- Group L: Patients with menstrual cycle between 20-24 were called Group L (Luteal phase)

SUMMARY:
The investigators aimed to investigate the effect of menstrual cycle phases on preoperative anxiety in women under general anesthesia.

DETAILED DESCRIPTION:
In preoperative period, preoperative anxiety is experienced in different degrees due to surgery and anesthesia. Preoperative anxiety is a condition that negatively affects anesthesia, surgery and postoperative recovery. It is reported that the incidence of preoperative anxiety in the western population is between 60% and 80%. In the pre-operative period, there are many causes of anxiety related to the patient's health and the concerns about the operation, uncertainty of the outcome, non-wake up after surgery, pain hearing and waking during surgery. It has been reported that anxiety increases direct blood pressure and changes pulse rate. It is stated that anxiety also affects the awakening criteria in postoperative period. This may cause hemodynamic instability in anesthesia applications.

Hormonal, physical and psychological fluctuations occur in women due to menstrual cycle. Therefore, it is reported that there is a strong relationship between the menstrual cycle and the person's emotional state. It is known that women feel good in the first phase of the cycle and they experience emotional, physical and behavioral disorders towards the end of the cycle. Studies have shown that anesthetic requirements, postoperative analgesic requirement and incidence of nausea vomiting may change with the phases of the cycle. Similarly, in the luteal phase of the cycle, it has been suggested that luteinizing hormones cause sensitization in opioid receptors and increase sensitivity to pain. In addition, depressive symptoms increase before menstruation. In this process, some women may have pre-menstrual dysphoric discomfort, irritability, mood swings, depression, flare, anger, restlessness, anorexia, sleep disturbance, and fatigue.

Our hypothesis is that preop anxiety will be higher in the surgeries planned in the luteal phase.

We aimed to investigate the effect of menstrual cycle phases on preoperative anxiety in women under general anesthesia.

Material Method Ethics Committee approval was obtained before the study. After the written consent of the patients were obtained, they started to the study. The study was planned as a randomized prospective study between February 2018 and February 2019.

The study groups were selected from patients who presented to the preop anesthesia polyclinic in elective conditions, septo-rinoplasty operation under general anesthesia. Assuming that there would be a 5-point difference in anxiety scores among the groups, it was decided to take 40 cases for each group with a 0.75 standard effect size, 80% power, and 5% error. Patients were randomly assigned to two groups of 40 patients. The patients were randomized by sequential addition to the groups determined in the order of their inclusion.

Study inclusion criteria: The study included 80 women with ASA I-II, aged 18 to 45 years, who were accepted to participate in the study, were smoking, did not use oral contraceptives, had no menstrual irregularity (regular 28 ± 2 days menstrual cycle).

Study exclusion criteria: In preop evaluation patients had difficulties in communication, amenorrhea, pregnancy, delirium, psychological illness, major depressive disorder, patients with a history of acute illness (such as in intensive care unit follow-up), which may affect cognitive function and daily life activities in the last 6 months, malignancy, acute renal failure, substance abuse and patients older than 45 years and male sex will be excluded from the study.

Groups:

Information about menstrual cycle patterns was obtained from all cases. The days of the menstrual cycle will be determined starting from counting the first day of the last cycle. Patients with menstrual cycle between 8-12 days were called Group F (Follicular phase). Patients with menstrual cycle between 20-24 were called Group L (Luteal phase). The follow-up of the cases and the recording of the measurements were performed by an anesthesiologist who did not know which group the cases were in.

Procedure to be Applied:

The sex, age, height and ASA scores of the patients were recorded preoperatively. The STAI instantaneous anxiety inventory, which measures situational anxiety in the preop unit, will be completed. In this form, there are 20 expressions, each is scored between the values of 1 to 4.

The total STAI score will be determined by subtracting the sum of the scores given to the expressions expressing positive emotions (1, 2, 5, 8, 10, 11, 15, 16, 19 and 20) from the sum of the scores given to the expressions expressing negative emotions (3, 4, 6, 7, 9, 12, 13, 14, 17 ve 18), then constant 50 number will be added to this value.

In preop unit and operation room, hemodynamic parameters (systolic, diastolic and mean arterial pressure (MAP), heart rate (HR) and peripheral oxygen saturation values preop at 15th, 10th, 5th, before induction, after induction at 1th and intubation at 1st, 5th and 15th minutes will be recorded.

Instead of patients who do not want to be included in the study or who are excluded from the study for any reason, according to the results of the power analysis, a targeted number of patients will be included in the study randomly.

ELIGIBILITY:
Inclusion Criteria:

* The study included 80 women with ASA I-II,
* Aged 18 to 45 years, who were accepted to participate in the study,
* were smoking,
* did not use oral contraceptives,
* had no menstrual irregularity (regular 28 ± 2 days menstrual cycle)

Exclusion Criteria:

* In preop evaluation patients had difficulties in communication,
* amenorrhea,
* pregnancy,
* delirium,
* psychological illness,
* major depressive disorder,
* patients with a history of acute illness (such as in intensive care unit follow-up),
* which may affect cognitive function and daily life activities in the last 6 months,
* malignancy,
* acute renal failure,
* substance abuse and patients older than 45 years and male sex will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study is performed on female gender with menstrual cycle.
Study Population: It will be operated for elective surgery, aged 18 to 45 years, who were accepted to participate in the study,
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety | 1 month
  Preoperative anxiety level will be measured by State-Trait Anxiety Inventory (STAI) form.

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yuzkat, Assist Prof, Study Chair — Yuzuncu Yil University
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)